CLINICAL TRIAL: NCT00831376
Title: A Proof of Concept Study to Evaluate the Trough Bronchoprotection Conferred by Chronic Dosing With Levosalbutamol and Racemic Salbutamol in Persistent Asthmatics
Brief Title: Trough Bronchoprotection Conferred by Levosalbutamol and Racemic Salbutamol
Acronym: NAI009
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, Brian J Lipworth, Professor, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NAI009
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Asthma
Keywords: Asthma; Genotype; Beta2adrenoreceptor; Levosalbutamol
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- levosalbutamol (Experimental): Patients will be asked to take two puffs four times a day for 2 weeks
  Interventions: Drug: levosalbutamol
- 2: racemic salbutamol (Active Comparator): Patients will be asked to take two puffs four times a day for 2 weeks
  Interventions: Drug: racemic salbutamol
- 3: Placebo (Placebo Comparator): Patients will be asked to take two puffs four times a day for 2 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: levosalbutamol — Patients will be asked to take two puffs four times a day for 2 weeks
  Arms: levosalbutamol
Drug: racemic salbutamol — Patients will be asked to take two puffs four times a day for 2 weeks
  Other Names: Ventolin
  Arms: 2: racemic salbutamol
Drug: placebo — Patients will be asked to take two puffs four times a day for 2 weeks
  Arms: 3: Placebo

SUMMARY:
The objective of this study is to compare the relative bronchoprotection (at trough) conferred by 2-week chronic dosing with levosalbutamol and racemic salbutamol in mild to moderate asthmatics. Patients will be preselected into two groups on the basis of their beta-2 adrenoreceptor polymorphisms. The investigators will evaluate if this has a differential effect on the bronchoprotection conferred by both formulations of salbutamol, as evidenced by a rebound in airway hyper-responsiveness, in order to determine whether any effect can be explained by the S enantiomer in the racemic formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Mild to moderate stable asthmatics on ≤ 2000μg BDP or equivalent, who are methacholine responsive PC20< 4 mg/ml
2. >1dd change in methacholine PC20 after the administration of racemic Salbutamol.
3. Male or female 18-65
4. Informed Consent
5. Ability to comply with the requirements of the protocol

Exclusion Criteria:

1. Severe asthmatics as defined by an FEV1≤ 60% or PEF variability > 30% or with continual daytime or nocturnal symptoms.
2. The use of oral corticosteroids within the last 3 months.
3. Recent respiratory tract infection (2 months).
4. Significant concomitant respiratory disease such as COPD, CF, ABPA, bronchiectasis and active pulmonary tuberculosis.
5. Any other clinically significant medical condition such as unstable angina, acute myocardial infarction in the preceding 3 months, recent TIA/ CVA, that may endanger the health or safety of the participant, or jeopardise the protocol.
6. Any significant abnormal laboratory result as deemed by the investigators
7. Pregnancy, planned pregnancy or lactation
8. Known or suspected contra-indication to any of the IMP's
9. Concomitant use of medicines (prescribed, over the counter or herbal) that may interfere with the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
methacholine challenge | before and after 2 week study period

SECONDARY OUTCOMES:
spirometry | before and after 2 week study period
nitric oxide levels | before and after 2 week study period
symptom scores | before and after 2 week study period
Bmax and Emax | before and after 2 week study period

CONTACTS AND LOCATIONS:
Overall Officials: Karine L Clearie, MBBS, MRCP, Principal Investigator — Asthma and Allergy Research Group; Brian J Lipworth, MBchB, Study Director — Asthma and Allergy Research Group
Locations (1):
- Asthma and Allergy Research Group, Dundee, Angus, United Kingdom

REFERENCES:
- [Result] Anderson WJ, Short PM, Williamson PA, Morrison AE, Palmer C, Tavendale R, Lipworth BJ. Proof-of-concept evaluation of trough airway hyper-responsiveness following regular racemic or levosalbutamol in genotype-stratified steroid-treated persistent asthmatic patients. Clin Sci (Lond). 2014 Jan 1;126(1):75-83. doi: 10.1042/CS20130213. PMID 23829494